CLINICAL TRIAL: NCT02639013
Title: Temporal Trend Analysis of Nurse's Knowledge and Practice Before and After Implementing an Educational Program Regarding Abdominal Compartment Syndrome
Brief Title: an Educational Program About Abdominal Compartment Syndrome
Acronym: Ghada
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Shalaby, lecturer in critical care nursing department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAH100
Record Dates: First submitted 2015-12-17; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Intraabdominal Hypertension
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ttransducer technique (Experimental): the nurses will measure intraabdominal pressure at each shift during the day by using transducer technique
  Interventions: Procedure: transducer technique

INTERVENTIONS:
Procedure: transducer technique — the nurses will receive the intervention ( the transducer method) to measure intraabdominal pressure intraabdominal hypertension and how to measure intraabdominal pressure in the third section
  Other Names: monitoring intraabdominal pressure

SUMMARY:
Early detection of intra-abdominal hypertension is essential to the prevention of abdominal compartment syndrome and requires close surveillance of intra-abdominal hypertension in patients at increased risk. intra-abdominal hypertension measurements are often taken by the bedside nurse, and in some cases, initiation of serial intra-abdominal hypertension monitoring is prompted by critical care nurses.

DETAILED DESCRIPTION:
Measurement of intra-abdominal pressure is simple, inexpensive, safe and accurate method in determining the presence of intra-abdominal hypertension. This measurement can guide patient management. Monitoring intra-abdominal pressure and abdominal per-fusion pressure.

for signs of abdominal compartment syndrome has become an inexpensive and useful diagnostics tool for identifying complications. An integrated approach to screening and monitoring for intra-abdominal hypertension may improve patient outcomes and decrease hospital costs. Due to the high incidence of intra-abdominal hypertension and abdominal compartment syndrome, it is essential for critical care nurses to regularly monitor intra-abdominal pressure and abdominal per-fusion pressure.

Critical care nurses have the ability to identify intra-abdominal hypertension and abdominal compartment syndrome, implement and evaluate management interventions. Nursing practice should be centered on evidence based practice guidelines . Nurses should provide a standard of care in managing patients who are at risk of intra-abdominal hypertension and abdominal compartment syndrome from pre hospital, emergency, operating room and intensive care areas

ELIGIBILITY:
Inclusion Criteria:

* all nurses that have more than one years experience in the trauma ,general and gastrointestinal ICU

Exclusion Criteria:

* nurses less than one year experience

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-04 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
improve nurses knowledge and practice about abdominal compartment syndrome | 6 months
  pretest and post questionaire will be used to evaluate the improvement in nurses knowledge and practice about abdominal compartment syndrome

SECONDARY OUTCOMES:
prevent abdominal compartment syndrome | 3 months
  measure inta-abdominal pressure correctly and continuously monitor signs of increased intrabdominal pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Sh Khalaf, Lecturer, Principal Investigator — Assuit university hospital
Locations (1):
- Faculty of Nursing, Egypt, Assuit, Egypt

REFERENCES:
- [Background] Newcombe J, Mathur M, Bahjri K, Ejike JC. Pediatric critical care nurses' experience with abdominal compartment syndrome. Ann Intensive Care. 2012 Jul 5;2 Suppl 1(Suppl 1):S6. doi: 10.1186/2110-5820-2-S1-S6. Epub 2012 Jul 5. PMID 22873422
- [Background] Hunt L, Frost SA, Hillman K, Newton PJ, Davidson PM. Management of intra-abdominal hypertension and abdominal compartment syndrome: a review. J Trauma Manag Outcomes. 2014 Feb 5;8(1):2. doi: 10.1186/1752-2897-8-2. PMID 24499574